CLINICAL TRIAL: NCT03594058
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Oral Solabegron Modified Release Tablets in the Treatment of Overactive Bladder (OAB) in Adult Female Subjects
Brief Title: A Study to Evaluate Once Daily Low Dose and High Dose Solabegron or Placebo Given for 12 Weeks to Treat Women With Symptoms of Overactive Bladder: Sudden Urge to Urinate, Frequent Urination Associated With Wetting Episodes (VEL-2001)
Acronym: VEL-2001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Velicept Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VEL-2001
Record Dates: First submitted 2018-07-09; First posted 2018-07-20 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2019-08

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; urinary conditions; urgency urinary incontinence; urgency; micturitions
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: This is a Phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel-group study. Eligible female subjects (N=1200) with symptoms of overactive bladder for at least 6 months will enter a 14-day single-blind Run-in Period. Subjects (N=375) who meet prespecified criteria based on data entered into an electronic diary over 3 days will be randomized 1:1:1 (125 subjects per arm) to receive solabegron modified release tablets, low dose or high dose, or matching placebo.
Who Masked: Participant, Investigator
Masking Description: Sponsor representatives Site monitors Data managers Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Solabegron modified release tablets low dose (Experimental)
  Interventions: Drug: Solabegron modified release tablets, low dose
- Solabegron modified release tablets high dose (Experimental)
  Interventions: Drug: Solabegron modified release tablets, high dose
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Solabegron modified release tablets, low dose — Solabegron modified release tablets low dose or high dose or matching placebo once daily for 12 weeks.
  Arms: Solabegron modified release tablets low dose
Drug: Solabegron modified release tablets, high dose — Solabegron modified release tablets low dose or high dose or matching placebo once daily for 12 weeks.
  Arms: Solabegron modified release tablets high dose
Drug: Matching Placebo — Solabegron modified release tablets low dose or high dose or matching placebo once daily for 12 weeks.
  Arms: Placebo Comparator

SUMMARY:
This is a Phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel-group study designed to evaluate the efficacy, safety, and tolerability of solabegron modified release low dose or high dose tablets, compared to matched placebo, administered once daily for 12 weeks to adult female subjects with overactive bladder symptoms (frequency, urgency, and predominantly urgency incontinence) for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult female subjects 18 to 80 years of age, with a ≥ 6-month history of symptoms of overactive bladder including: frequency, urgency, urgency urinary incontinence, and mixed incontinence. Subjects must provide written informed consent and either be of non-childbearing potential or of childbearing potential meeting specific criteria (e.g., negative pregnancy test, sexual inactivity, acceptable methods of birth control, and use of hormonal contraceptives).

Exclusion Criteria:

* Subjects must have no history of pelvic or bladder disease, e.g., uterine prolapse, malignancy, prior surgery, or treatment with botulinum toxin.
* Diabetes insipidus or poorly controlled Type 1 or Type 2 diabetes mellitus
* Cardiac conditions:
* prior cardiovascular events or procedures within 6 months of screening
* congestive heart failure
* abnormal ECG findings, including ECG QT correction interval (QTc) > 470 msec at the Screening Visit
* systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg, or heart rate > 100 beats per minute
* Abnormal tests of liver function
* History of prior infection due to HIV or hepatitis B or hepatitis C virus
* Allergy or hypersensitivity to solabegron or mirabegron
* Women of childbearing potential: breastfeeding, pregnant, or actively trying to become pregnant
* Participation in a trial of an investigational or marketed drug ≤ 30 days prior to the Screening Visit or in any clinical trial of an investigational drug that may affect urinary function within 3 months prior to Screening Visit.
* Inability to read, understand, or complete study-related materials

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1413 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in mean number of micturitions per 24 hours at Week 12 | Micturtions will be assessed prior to randomization and at Week 12 (Visit 6).
  Micturition events will be recorded by subjects in an eDiary using a smartphone device during 3-day diary periods prior to randomization and at 12 weeks.

SECONDARY OUTCOMES:
Urinary Incontinence (1) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in mean number of urgency urinary incontinence episodes per 24 hours
Urinary Incontinence (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage change from Baseline in mean number of urgency urinary incontinence episodes per 24 hours
Urinary Incontinence (3) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Proportion of subjects with no episodes of urgency urinary incontinence per 24 hours
Urinary Incontinence (4) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Proportion of subjects with no episodes of urinary incontinence (urgency and non-urgency) per 24 hours
Urinary Incontinence (5) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in total urinary incontinence episodes (urgency and non-urgency) per 24 hours
Micturitions (1) | Prior to Randomization (Baseline) and at Weeks 4 and 8
  Change from Baseline in mean number of micturitions per 24 hours
Micturitions (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage change from Baseline in mean number of micturitions per 24 hours
Micturitions (3) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage of subjects with < 8 micturitions per 24 hours
Micturitions (4) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in mean number of nocturnal voids per 24 hours
Urine Void Volume (1) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in average void volume over 24 hours
Urine Void Volume (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage change from Baseline in average void volume over 24 hours
Urine Void Volume (3) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in maximum individual void volume over 24 hours
Urine Void Volume (4) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage change from Baseline in maximum individual void volume over 24 hours
Urgency (1) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Proportion of subjects with urges with a mean grade of 3 of 4 per 24 hours
Urgency (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in mean urgency assessments per 24 hours associated with micturitions or incontinence
Patient Reported Outcomes (1) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Patient Perception of Bladder Control. This patient-reported questionnaire assesses the patient's perception of current urinary problems, where higher score (on a scale of 1 to 6) indicates more severe problems.
Patient Reported Outcomes (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in Symptom Bother Score (Overactive Bladder Questionnaire [OAB-q] short form). The OAB-q short form is completed as a 4-week recall where a higher score (on a scale of 1 to 6) indicates greater symptoms.
Patient Reported Outcomes (3) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in health-related quality of life (Overactive Bladder Questionnaire [OAB-q] short form). The OAB-q short form is completed as a 4-week recall where a higher score (on a scale of 1 to 6) indicates worse health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (66):
- United States (66):
  - Velicept Investigative Site - Birmingham, Birmingham, Alabama
  - Velicept Investigative Site - Guntersville, Guntersville, Alabama
  - Velicept Investigative Site - Saraland, Saraland, Alabama
  - Velicept Investigative Site - Tucson, Tucson, Arizona
  - Velicept Investigative Site - Lincoln, Lincoln, California
  - Velicept Investigative Site - North Hollywood, North Hollywood, California
  - Velicept Investigative Site - Sacramento, Sacramento, California
  - Velicept Investigative Site - San Diego, San Diego, California
  - Velicept Investigative Site - Spring Valley, Spring Valley, California
  - Velicept Investigative Site - Upland, Upland, California
  - Velicept Investigative Site - Aurora, Aurora, Colorado
  - Velicept Investigative Site - Englewood, Englewood, Colorado
  - Velicept Investigative Site - New London, New London, Connecticut
  - Velicept Investigative Site - Aventura, Aventura, Florida
  - Velicept Investigative Site - Doral(2), Doral, Florida
  - Velicept Investigative Site - Doral, Doral, Florida
  - Velicept Investigative Site - Edgewater, Edgewater, Florida
  - Velicept Investigative Site - Hialeah, Hialeah, Florida
  - Velicept Investigative Site - Hollywood, Hollywood, Florida
  - Velicept Investigative Site - Lauderdale Lakes, Lauderdale Lakes, Florida
  - Velicept Investigative Site - Miami, Miami, Florida
  - Velicept Investigative Site - Miami Springs, Miami Springs, Florida
  - Velicept Investigative Site - New Port Richey, New Port Richey, Florida
  - Velicept Investigative Site - Palm Harbor, Palm Harbor, Florida
  - Velicept Investigative Site - Pompano Beach, Pompano Beach, Florida
  - Velicept Investigative Site - Tampa, Tampa, Florida
  - Velicept Investigative Site - West Palm Beach, West Palm Beach, Florida
  - Velicept Investigative Site - Atlanta, Atlanta, Georgia
  - Velicept Investigative Site - Snellville, Snellville, Georgia
  - Velicept Investigative Site - Crowley, Crowley, Louisiana
  - Velicept Investigative Site - Metairie, Metairie, Louisiana
  - Velicept Investigative Site - Brighton, Brighton, Massachusetts
  - Velicept Investigative Site - North Dartmouth, North Dartmouth, Massachusetts
  - Velicept Investigative Site - Saginaw, Saginaw, Michigan
  - Velicept Investigative Site - Biloxi, Biloxi, Mississippi
  - Velicept Investigative Site - Olive Branch, Olive Branch, Mississippi
  - Velicept Investigative Site - La Vista, La Vista, Nebraska
  - Velicept Investigative Site - Las Vegas, Las Vegas, Nevada
  - Velicept Investigative Site - Edison, Edison, New Jersey
  - Velicept Investigative Site - Raleigh, Raleigh, North Carolina
  - Velicept Investigative Site - Fargo, Fargo, North Dakota
  - Velicept Investigative Site - Dayton, Dayton, Ohio
  - Velicept Investigative Site - Mustang, Mustang, Oklahoma
  - Velicept Investigative Site - Oklahoma City, Oklahoma City, Oklahoma
  - Velicept Investigative Site - Gresham, Gresham, Oregon
  - Velicept Investigative Site - Lansdale, Lansdale, Pennsylvania
  - Velicept Investigative Site - East Providence, East Providence, Rhode Island
  - Velicept Investigative Site - Lincoln, Lincoln, Rhode Island
  - Velicept Investigative Site - Charleston, Charleston, South Carolina
  - Velicept Investigative Site - Fort Mill, Fort Mill, South Carolina
  - Velicept Investigative Site - Spartanburg, Spartanburg, South Carolina
  - Velicept Investigative Site - Chattanooga, Chattanooga, Tennessee
  - Velicept Investigative Site - Jackson, Jackson, Tennessee
  - Velicept Investigative Site - Knoxville, Knoxville, Tennessee
  - Velicept Investigative Site - Austin, Austin, Texas
  - Velicept Investigative Site - Bryan, Bryan, Texas
  - Velicept Investigative Site - Carrollton, Carrollton, Texas
  - Velicept Investigative Site - Dallas, Dallas, Texas
  - Velicept Investigative Site - Fort Worth, Fort Worth, Texas
  - Velicept Investigative Site - Georgetown, Georgetown, Texas
  - Velicept Investigative Site - Houston, Houston, Texas
  - Velicept Investigative Site - Plano(1), Plano, Texas
  - Velicept Investigative Site - Plano(2), Plano, Texas
  - Velicept Investigative Site - San Angelo, San Angelo, Texas
  - Velicept Investigative Site - San Antonio, San Antonio, Texas
  - Velicept Investigative Site - Sugar Land, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohlstein EH, von Keitz A, Michel MC. A multicenter, double-blind, randomized, placebo-controlled trial of the beta3-adrenoceptor agonist solabegron for overactive bladder. Eur Urol. 2012 Nov;62(5):834-40. doi: 10.1016/j.eururo.2012.05.053. Epub 2012 Jun 5. PMID 22695239